CLINICAL TRIAL: NCT00803348
Title: The Secret Recipe for Femoral Nerve Blockade After Total Knee Arthroplasty: A Randomized, Placebo-controlled, Double-blind Trial
Brief Title: Continuous Femoral Nerve Blockade and Readiness to Discharge Following Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 08-0895-B
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Last update posted 2012-04-26 (Estimated); Status verified 2010-01

CONDITIONS: Knee Arthroplasty
Keywords: continuous femoral nerve blockade; knee arthroplasty; knee replacement; regional anesthesia; readiness to discharge; Femoral nerve blockade for total knee arthroplasty

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Initial Bolus dose of 0.2% ropivicaine followed by 0.2% ropivicaine infusion until day 2 post-op
  Interventions: Drug: Bolus of 0.2% ropivicaine 20 mls followed by 0.2% ropivicaine at an infusion rate of 5mls/hr until 0600 on postoperative day 2
- 2 (Experimental): Initial Bolus dose of 0.2% ropivicaine followed by 0.1% ropivicaine infusion until day 2 post-op
  Interventions: Drug: Bolus of 0.2% ropivicaine 20 mls followed by 0.1% ropivicaine at an infusion rate of 10mls/hr until 0600 on post-operative day 2
- 3 (Placebo Comparator): Initial Bolus dose of 0.375% ropivicaine followed by saline infusion until day 2 post-op
  Interventions: Drug: Saline control

INTERVENTIONS:
Drug: Bolus of 0.2% ropivicaine 20 mls followed by 0.2% ropivicaine at an infusion rate of 5mls/hr until 0600 on postoperative day 2 — Initial bolus of 0.2% ropivicaine 20 mls into the femoral catheter followed by 0.2% ropivicaine at an infusion rate of 5mls/hr with patient controlled boluses of 5ml available every 30 mins, until 0600 on the morning of postoperative day 2
  Arms: 1
Drug: Bolus of 0.2% ropivicaine 20 mls followed by 0.1% ropivicaine at an infusion rate of 10mls/hr until 0600 on post-operative day 2 — Initial bolus of 0.2% ropivicaine 20 mls into the femoral catheter followed by 0.1% ropivicaine at an infusion rate of 10mls/hr with patient controlled boluses of 10mls available every 30 mins, until 0600 on the morning of postoperative day 2
  Arms: 2
Drug: Saline control — Bolus of 0.375% ropivicaine 30 mls followed by saline infusion until 0600 on postoperative day 2
  Arms: 3

SUMMARY:
Patients undergoing total knee arthroscopy (knee replacement) surgery usually receive a femoral nerve block as part of their anesthetic care. Some centers administer the block with a single shot of local anesthetic, which wears off several hours after surgery. Other centers administer the block with a single shot followed by continuous infusion of local anesthetic, typically for 2 to 5 days after surgery. The latter method, though good for pain control, may result in decreased mobility (while the anesthetic is still active), longer hospital stays, and greater risk of falls.

This study will see if using a lower concentration of local anesthetic for the continuous femoral nerve block or only the initial single-shot dose will result in increased mobility and shorter hospital stays.

ELIGIBILITY:
Inclusion Criteria:

1. ASA physical status I-III
2. 18-85 years of age, inclusive
3. Able to communicate in English sufficiently to participate in the study
4. Able to walk 30 metres without stopping prior to surgery

Exclusion Criteria:

1. Intended discharge to in-patient rehabilitation facility
2. Patient refusal of FNB or spinal anesthetic or sciatic nerve block
3. Contraindications to peripheral nerve block (e.g. allergy to local anesthetics, refusal)
4. Significant peripheral neuropathy or neurological disorder affecting the lower extremity
5. Contraindication to a component of multi-modal analgesia
6. Pregnancy
7. History of use of over 30mg oxycodone or equivalent per day (institutional threshold for acute pain service consultation pre-operatively)
8. History of significant cognitive or psychiatric condition that may affect patient assessment
9. Inability to provide informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2009-05; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Time to readiness to discharge from hospital | Twice daily until discharge

SECONDARY OUTCOMES:
Quadriceps strength, knee flexion, walking distance, pain, patient satisfaction, opioid consumption, adverse events, incidence of falls, volume of local anesthetic administered, block success, discharge date, functional recovery | Up to Month 6 post-operative

CONTACTS AND LOCATIONS:
Overall Officials: Richard Brull, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Albrecht E, Morfey D, Chan V, Gandhi R, Koshkin A, Chin KJ, Robinson S, Frascarolo P, Brull R. Single-injection or continuous femoral nerve block for total knee arthroplasty? Clin Orthop Relat Res. 2014 May;472(5):1384-93. doi: 10.1007/s11999-013-3192-3. PMID 23928707